CLINICAL TRIAL: NCT00182754
Title: An Exploratory, Randomized, Placebo-Controlled Trial of Depot Octreotide (Sandostatin LARDepot) for Symptomatic Ascites in Cancer Patients
Brief Title: Octreotide in Treating Patients With Cancer-Related Malignant Ascites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-N04C2; NCI-2009-00647 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000440922 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; malignant ascites
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive octreotide subcutaneously (SC) once on day 1.
  Interventions: Drug: octreotide acetate
- Arm II (Placebo Comparator): Patients receive placebo SC once on day 1.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: octreotide acetate — Given subcutaneously
  Arms: Arm I
Other: placebo — Given subcutaneously
  Arms: Arm II

SUMMARY:
RATIONALE: Octreotide may be an effective treatment for malignant ascites. It is not yet known whether octreotide is more effective than a placebo in treating malignant ascites.

PURPOSE: This randomized phase III trial is studying octreotide to see how well it works compared to placebo in treating patients with cancer-related malignant ascites.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of octreotide vs placebo, in terms of extending the time-to-paracentesis, in patients with cancer-related symptomatic malignant ascites.

Secondary

* Compare the number of paracenteses in patients treated with these drugs.
* Determine the toxicity of octreotide in these patients.
* Compare the quality of life of patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to anticipated ongoing chemotherapy (yes vs no), frequency of prior paracentesis (never vs other), and prior chemotherapy (never vs only first-line chemotherapy vs second-line chemotherapy vs other). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive octreotide subcutaneously (SC) once on day 1.
* Arm II: Patients receive placebo SC once on day 1. In both arms, treatment with intramuscular octreotide or placebo repeats monthly for up to 2 years in the absence of unacceptable toxicity.

Quality of life is assessed at baseline, 2 weeks, and then monthly for up to 2 years during study treatment.

After completion of study treatment, patients are followed every 6 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cancer
* Diagnosis of malignant ascites, as determined by the treating oncologist

  * Positive cytology not required
  * Patient is symptomatic and views ascites as a problem
* No lymphoma or lymphomatous ascites
* Planning therapeutic paracentesis ≤ 3 days after study entry OR completed therapeutic paracentesis 2 days before study entry

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* At least 4 weeks

Hematopoietic

* Not at high risk of bleeding from a procedure

Hepatic

* No known cirrhosis or portal hypertension

Renal

* No known history of chronic renal failure, defined as creatinine ≥ 2 times upper limit of normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Prior cholecystitis allowed provided patient underwent cholecystectomy
* No uncontrolled diabetes mellitus
* No known allergy to octreotide
* No known allergy to latex
* No medical condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent bevacizumab

Chemotherapy

* No concurrent intraperitoneal chemotherapy
* No concurrent first-line chemotherapy for any cancer except pancreatic cancer

  * Concurrent second-line chemotherapy or later-line chemotherapy allowed

Endocrine therapy

* No other concurrent octreotide

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent therapeutic warfarin

  * Concurrent prophylactic warfarin at a dose of 1 mg/day allowed
* No other concurrent treatment for ascites except paracentesis or ongoing diuretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-10; Primary Completion 2009-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (122):
- United States (122):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fergus Falls, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive 30 mg octreotide subcutaneously (SC) intramuscularly once on day 1. octreotide acetate: Given subcutaneously
- Arm II: Patients receive 2 milliliters placebo (0.9% sodium chloride) SC once on day 1. placebo: Given subcutaneously
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 90] | 69 [40 to 88] | 63 [40 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Paracentesis
Description: Kaplan Meier curves will be constructed for each group; patients lost to follow up will be censored. A log rank test will be used to compare groups. We will adjust for the volume of fluid withdrawn at paracentesis and for change in abdominal circumference between baseline and the next procedure because a patient may require an extra paracentesis if only a small volume is withdrawn at baseline.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 16 | 17
days | 28 [4 to 45] | 14 [4 to 28]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.17, Log Rank

2. Secondary Outcome: Number of Paracenteses
Description: We will compare the number of paracenteses between groups. Parametric or nonparametric testing will be used as appropriate.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: number of paracenteses per patient
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 16 | 17
number of paracenteses per patient | 0.5 [0 to 4] | 1 [0 to 4]

3. Secondary Outcome: Average Quality-of-life
Description: Quality of life will be recorded and analyzed in a descriptive, exploratory fashion. We acknowledge that this study will represent the first to attempt a prospective assessment of quality of life in patients with symptomatic ascites. The underlying hypothesis of this quality of life assessment is that patients who are receiving octreotide will enjoy a better quality of life compared to patients who receive placebo. Quality of life scores from the CLDQ will be summed for all patients on a monthly basis. Again we anticipate high patient drop out rates over time within these two cohorts. With due diligence, we will attempt to ascertain the reason for each patient drop out, and appropriate imputation techniques will be employed for each.Quantified as: 1='All of the time' 2='Most of the time' 3='A good bit of the time' 4='Some of the time' 5='A little bit of the time' 6='Hardly any of the time' 7='None of the time' 0='Missing';
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: QOL score
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 10 | 15
QOL score
  abdominal bloating | 4 [1 to 6] | 3 [1 to 6]
  shortness of breath | 4 [3 to 7] | 3 [1 to 6]
  abdominal discomfort | 4.5 [2 to 5] | 2 [1 to 6]

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17
Other Adverse Events (participants affected / at risk) | 16/16 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=16) | Arm II (N=17)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=16) | Arm II (N=17)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (20) | 12 (14)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (10) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 4 (14) | 5 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Proctitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 3 (4) | 2 (2)
Injection site reaction (General disorders) | 1 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 0 (0)
Platelet count decreased (Investigations) | 1 (4) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vascular disorder (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes